CLINICAL TRIAL: NCT05294562
Title: China Post-Market Clinical Follow-up of FACILLE®
Status: Completed | Type: Observational
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PMCF-FE01
Record Dates: First submitted 2022-03-10; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Dermal Filler; Hyaluronic Acid; Nasolabial Fold

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The results showed that subjects tolerated the Sodium Hyaluronate Gel for Injection (FACILLE®) well, with no systemic AEs, SAEs, and unanticipated AEs and associated with high satisfaction and self-evaluated effectiveness. Nearly half of the subjects maintained correction for 12 months and were satisfied with the product 3 years after the first injection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older of male or female;
* Have used or plan to use FACILLE® Sodium Hyaluronate Gel for Injection;
* Agree to participate and comply with the follow-up schedule of this study.

Exclusion Criteria:

* With a history of hypersensitivity or allergy to hyaluronic acid or any component of the device;
* Other circumstances were judged to be unsuitable for participating in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Institution of Medical Cosmetology
Sampling Method: Non-Probability Sample
Enrollment: 1552 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Adverse events reported during the study period | 36 months
  The safety assessment was based on reports of adverse events, defined as any unwanted events whether it was thought to be related to the study drugs or not, were recorded during each follow up and at any time the patient reported an event to the investigator during the study period.

SECONDARY OUTCOMES:
Subjects self-evaluating satisfaction | 2 weeks, 1, 3, 6, 12, 18, 24, 30 and 36 months post-injection
  Patients rate their treatment satisfaction based on highly satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied.
Subjects self-evaluating effectiveness | 2 weeks, 1, 3, 6, 12, 18, 24, 30 and 36 months post-injection
  Patients rate their effectiveness based on effective and ineffective.